CLINICAL TRIAL: NCT04831541
Title: 68Ga-PSMA-11 PET/CT in Patients With Various Types of Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director, Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian6
Record Dates: First submitted 2020-09-05; First posted 2021-04-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer; Positron-Emission Tomography
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA-11 (Experimental): Each subject receive a single intravenous injection of 68Ga-PSMA-11, and undergo PET/CT imaging within the specificed time.
  Interventions: Drug: 68Ga-PSMA-11

INTERVENTIONS:
Drug: 68Ga-PSMA-11 — Each subject receive a single intravenous injection of 68Ga-PSMA-11, and undergo PET/CT imaging within the specificed time.
  Other Names: Diagnostic Test: PET/CT scan

SUMMARY:
To evaluate the potential usefulness of 68Ga-PSMA-11 positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions, efficacy assessment and recurrence monitoring in various types of cancer.

DETAILED DESCRIPTION:
Subjects with various types of cancer underwent 68Ga-PSMA-11 PET/CT either for an initial assessment or for recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 68Ga-PSMA-11 PET/CT were calculated.

ELIGIBILITY:
Inclusion Criteria:

(i) adult population (aged 18 years or order); (ii) patients with suspected or new diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report); (iii) patients who had scheduled 68Ga-PSMA-11 PET/CT scan; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

(i) patients with pregnancy; (ii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of 68Ga-PSMA-11 for each target lesion of subject or suspected primary tumor or/and metastasis.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity and accuracy of 68Ga-PSMA-11 PET/CT were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No